CLINICAL TRIAL: NCT00617279
Title: Comparison of Primary Patency Between GORE PROPATEN Vascular Graft and Disadvantaged Autologous Vein Graft For Below-Knee Arterial Bypass (PRODIGY Study)
Brief Title: GORE PROPATEN Vascular Graft vs. Disadvantaged Autologous Vein Graft
Acronym: PRODIGY
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study terminated due to low enrollment
Sponsor: W.L.Gore & Associates (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PPT 07-05
Record Dates: First submitted 2007-12-18; First posted 2008-02-18 (Estimated); Results first posted 2012-01-12 (Estimated); Last update posted 2012-01-12 (Estimated); Status verified 2011-12

CONDITIONS: Peripheral Arterial Occlusive Disease
MeSH Terms: conditions — Peripheral Arterial Occlusive Disease 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- GORE PROPATEN Vascular Graft: (Active Comparator)
  Interventions: Device: GORE PROPATEN Vascular Graft
- Disadvantaged Autologous Vein Graft (Active Comparator)
  Interventions: Procedure: Disadvantaged Autologous Vein Graft

INTERVENTIONS:
Device: GORE PROPATEN Vascular Graft — Arterial Occlusion Bypass
  Arms: GORE PROPATEN Vascular Graft:
Procedure: Disadvantaged Autologous Vein Graft — Arterial Occlusion Bypass
  Arms: Disadvantaged Autologous Vein Graft

SUMMARY:
The primary patency of the GORE PROPATEN Vascular Graft is equivalent to or better than disadvantaged autologous vein graft in an infragenicular peripheral bypass application at 12 months.

DETAILED DESCRIPTION:
Primary patency is defined as hemodynamic evidence of blood flow through an open graft that has maintained uninterrupted patency and has not previously undergone a revision to restore blood flow. A disadvantaged autologous vein is defined as meeting at least one of the two following criteria: (1) Any autologous vein(s) other than greater saphenous vein deemed usable by the Investigator; (2) Usable ipsilateral or contralateral autologous greater saphenous vein that meets any of the following criteria: (a) Diameter of less than or equal to 3.0 mm; (b) Inadequate length requiring splicing; (c) Poor quality vein that is either sclerotic or phlebitic.

ELIGIBILITY:
Inclusion Criteria:

1. Patient requires below-knee bypass secondary to severe claudication, rest pain or tissue loss due to peripheral arterial occlusive disease.
2. Patient meets the disadvantaged autologous vein criteria described in Section 4.1.
3. Patient has a post-operative life expectancy greater than one year.
4. Patient is at least 21 years of age.
5. Patient is able to comply with all study requirements and be available for follow-up visits at 1, 6, 12, 24 and 36-months post-procedure.
6. Patient is willing and able to provide written, informed consent.

Exclusion Criteria:

1. Patient has had a previous instance of Heparin Induced Thrombocytopenia type 2 (HIT-2) or has known hypersensitivity to heparin.
2. Patient requires an infragenicular bypass for reasons other than peripheral arterial occlusive disease.
3. Patient requires sequential extremity revascularizations or other procedures that require use of additional vascular grafts.
4. Patient is in need of, or is scheduled for, a cardiac surgical procedure or a different vascular surgical procedure within 30 days of study procedure. However, inflow procedures that facilitate the bypass are permitted, as long as they are not performed at the same sitting as the bypass procedure.
5. Patient has been previously randomized for this study.
6. Patient has active infection in the region of graft placement.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2007-12; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard F. Neville, MD, Principal Investigator — Georgetown University Hospital; Jennifer Recknor, Ph.D., Study Director — W.L.Gore & Associates
Locations (17):
- United States (17):
  - University Of Alabama Medical Center, Birmingham, Alabama
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - Emory University School of Medicine, Atlanta, Georgia
  - Medical Center of Central Georgia, Macon, Georgia
  - University of Chicago, Chicago, Illinois
  - Vascular Specialty Associates, Baton Rouge, Louisiana
  - University of Maryland Medical Center, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Albany Medical Center, Albany, New York
  - Stonybrook University Medical Center, Stony Brook, New York
  - Montifiore Medical Center, The Bronx, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Greenville Hospital System, Greenville, South Carolina
  - University of Tennessee medical Center, Knoxville, Tennessee
  - The Methodist Hospital System, Houston, Texas
  - Peripheral Vascular Associates, San Antonio, Texas
  - Sentara Norfolk Hospital, Norfolk, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients requiring below-knee bypass secondary to severe claudication, rest pain or tissue loss due to peripheral arterial occlusive disease were recruited. Recruitment commenced December 2007 and was terminated by the Sponsor January 2010 due to slow enrollment. Investigative site locations included university hospitals and other medical clinics.
Groups:
- GORE PROPATEN Vascular Graft:: Patients receiving the GORE PROPATEN Vascular Graft in a below-knee bypass due to severe claudication (pain, tension, and weakness in the legs), rest pain or tissue loss due to peripheral arterial occlusive disease.
- Disadvantaged Autologous Vein Graft: Patients receiving Disadvantaged Autologous Vein Graft in a below-knee bypass due to severe claudication (pain, tension, and weakness in the legs), rest pain or tissue loss due to peripheral arterial occlusive disease. 'Disadvantaged Autologous Vein Graft' was defined in the study as meeting one of two criteria: (1) Any autologous vein(s) other than greater saphenous vein deemed usable by the Investigator (and/or) (2) Usable ipsilateral or contralateral autologous greater saphenous vein that is either less than or equal to 3.0 mm in diameter, of inadequate length (requires vein splicing), or of poor quality vein (sclerotic or phlebitic).
Period: Overall Study
Arm/Group | GORE PROPATEN Vascular Graft: | Disadvantaged Autologous Vein Graft
Started | 14 | 17
Completed | 0 | 0
Not Completed | 14 | 17
Not completed — Study terminated by Sponsor | 10 | 15
Not completed — Graft abandonment | 2 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Death | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GORE PROPATEN Vascular Graft: | Disadvantaged Autologous Vein Graft | Total
Number analyzed (Participants) | 14 | 17 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 7 | 14
  >=65 years | 7 | 10 | 17
Age Continuous [Mean (Standard Deviation); unit: years] | 65 (10) | 68 (8) | 67 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 7 | 12 | 19
Region of Enrollment [Number; unit: participants]
  United States | 14 | 17 | 31

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Primary Patency at 12 Months Post-procedure
Description: Primary patency is defined as hemodynamic evidence of blood flow through an open graft that has maintained uninterrupted patency and has not previously undergone a revision to restore blood flow.
Time Frame: 12 months
Population: The number of patients analyzed at 12 months post-procedure does not equal the number of patients originally enrolled into the study. This is due to the fact that many enrolled patients did not have their 12 month follow-up visit prior to the termination of the study.
Measure: Number; unit: Participants
Arm/Group | GORE PROPATEN Vascular Graft: | Disadvantaged Autologous Vein Graft
Number analyzed (Participants) | 6 | 7
Participants
  Patent | 2 | 3
  Lost Patency | 4 | 4

2. Secondary Outcome: Number of Patients With Primary Patency at One Month Post-procedure
Description: as for outcome 1
Time Frame: One month
Population: The number of patients analyzed at 1 month post-procedure does not equal the number of patients originally enrolled into the study. This is due to the fact that a number of enrolled patients did not have their 1 month follow-up visit (or failed to attend their 1 month visit) prior to the termination of the study.
Measure: Number; unit: Participants
Arm/Group | GORE PROPATEN Vascular Graft: | Disadvantaged Autologous Vein Graft
Number analyzed (Participants) | 10 | 8
Participants
  Patent | 8 | 5
  Lost Patency | 2 | 3

3. Primary Outcome: Major Adverse Event Occurrences Through One Month Post-procedure
Description: The number of Major Adverse Event occurrences through one month post-procedure. A major adverse event requires significant therapy, including unplanned increase in the level of care, permanent sequelae, hospitalization, or death. This outcome measure presents the number of Major Adverse Event occurrences (i.e. - one patient could have multiple occurrences), and differs from the Serious Adverse Events reporting measure, which presents the number of patients that have been affected by a Serious Adverse Event.
Time Frame: one month post-index procedure
Measure: Number; unit: Events
Arm/Group | GORE PROPATEN Vascular Graft: | Disadvantaged Autologous Vein Graft
Number analyzed (Participants) | 14 | 17
Events | 4 | 5

4. Secondary Outcome: Number of Patients With Primary Patency at 6 Months Post-procedure
Description: as for outcome 1
Time Frame: 6 months
Population: The number of patients analyzed at 6 months post-procedure does not equal the number of patients originally enrolled into the study. This is due to the fact that a number of enrolled patients did not have their 6 month follow-up visit (or failed to attend their 6 month visit) prior to the termination of the study.
Measure: Number; unit: Participants
Arm/Group | GORE PROPATEN Vascular Graft: | Disadvantaged Autologous Vein Graft
Number analyzed (Participants) | 8 | 9
Participants
  Patent | 5 | 5
  Lost patency | 3 | 4

5. Secondary Outcome: Number of Patients With Assisted Primary Patency at One Month Post-procedure
Description: Assisted primary patency is defined as hemodynamic evidence of blood flow through an open graft that has previously undergone revision(s) within the graft to restore blood flow prior to occlusion. The number of patients analyzed at 1 month post-procedure does not equal the number of patients originally enrolled into the study. This is due to the fact that a number of enrolled patients did not have their 1 month follow-up visit (or failed to attend their 1 month visit) prior to the termination of the study.
Time Frame: One month
Measure: Number; unit: Participants
Arm/Group | GORE PROPATEN Vascular Graft: | Disadvantaged Autologous Vein Graft
Number analyzed (Participants) | 8 | 10
Participants
  Patency | 5 | 8
  Lost Patency | 3 | 2

6. Secondary Outcome: Number of Patients With Assisted Primary Patency at 6 Months Post-procedure
Description: Assisted primary patency is defined as hemodynamic evidence of blood flow through an open graft that has previously undergone revision(s) within the graft to restore blood flow prior to occlusion.
Time Frame: 6 months
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | GORE PROPATEN Vascular Graft: | Disadvantaged Autologous Vein Graft
Number analyzed (Participants) | 8 | 8
Participants
  Patent | 5 | 5
  Lost patency | 3 | 3

7. Secondary Outcome: Number of Patients With Assisted Primary Patency at 12 Months Post-procedure
Description: as for outcome 6
Time Frame: 12 months
Population: The number of patients analyzed at 12 months post-procedure does not equal the number of patients originally enrolled into the study. This is due to the fact that a number of enrolled patients did not have their 12 month follow-up visit (or failed to attend their 12 month visit) prior to the termination of the study.
Measure: Number; unit: Participants
Arm/Group | GORE PROPATEN Vascular Graft: | Disadvantaged Autologous Vein Graft
Number analyzed (Participants) | 6 | 6
Participants
  Patent | 2 | 3
  Lost patency | 4 | 3

8. Secondary Outcome: Number of Patients With Secondary Patency at One Month
Description: Secondary patency is defined as hemodynamic evidence of blood flow through an open graft that has previously undergone revision(s) to restore blood flow after occlusion.
Time Frame: One month
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | GORE PROPATEN Vascular Graft: | Disadvantaged Autologous Vein Graft
Number analyzed (Participants) | 10 | 8
Participants
  Patent | 8 | 5
  Lost patency | 2 | 3

9. Secondary Outcome: Number of Patients With Secondary Patency at 6 Months
Description: as for outcome 8
Time Frame: 6 months
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | GORE PROPATEN Vascular Graft: | Disadvantaged Autologous Vein Graft
Number analyzed (Participants) | 7 | 8
Participants
  Patency | 5 | 5
  Lost patency | 2 | 3

10. Secondary Outcome: Number of Patients With Secondary Patency at 12 Months
Description: as for outcome 8
Time Frame: 12 months
Population: as for outcome 7
Measure: Number; unit: Participants
Arm/Group | GORE PROPATEN Vascular Graft: | Disadvantaged Autologous Vein Graft
Number analyzed (Participants) | 4 | 6
Participants
  Patent | 2 | 3
  Lost patency | 2 | 3

11. Secondary Outcome: Number of Patients With Limb Salvage (no Major Amputations) at One Month Post-procedure
Description: Limb salvage is defined as relief from symptoms sufficient to prevent major amputation. An amputation is considered to be major when there is surgical removal of a portion of the study leg that would preclude standing and walking without a prosthesis.
Time Frame: One month
Measure: Number; unit: Participants
Arm/Group | GORE PROPATEN Vascular Graft: | Disadvantaged Autologous Vein Graft
Number analyzed (Participants) | 14 | 17
Participants
  Limb salvaged | 13 | 17
  Limb not salvaged | 1 | 0

12. Secondary Outcome: Number of Patients With Limb Salvage (no Major Amputations) at 6 Months Post-procedure
Description: as for outcome 11
Time Frame: 6 months
Measure: Number; unit: Participants
Arm/Group | GORE PROPATEN Vascular Graft: | Disadvantaged Autologous Vein Graft
Number analyzed (Participants) | 14 | 17
Participants
  Limb salvaged | 13 | 17
  Limb not salvaged | 1 | 0

13. Secondary Outcome: Number of Patients With Limb Salvage (no Major Amputations) at 12 Months Post-procedure
Description: as for outcome 11
Time Frame: 12 months
Measure: Number; unit: Participants
Arm/Group | GORE PROPATEN Vascular Graft: | Disadvantaged Autologous Vein Graft
Number analyzed (Participants) | 14 | 17
Participants
  Limb salvaged | 13 | 17
  Limb not salvaged | 1 | 0

14. Secondary Outcome: Patients Experiencing Major Adverse Events Through 6 Months Post-procedure
Description: A major adverse event requires significant therapy, including unplanned increase in the level of care, permanent sequelae, hospitalization, or death.
Time Frame: 6 months
Measure: Number; unit: Participants
Arm/Group | GORE PROPATEN Vascular Graft: | Disadvantaged Autologous Vein Graft
Number analyzed (Participants) | 14 | 17
Participants
  Major Adverse Event occurred | 3 | 2
  Major Adverse Event did not occur | 11 | 15

15. Secondary Outcome: Patients Experiencing Major Adverse Events Through 12 Months Post-procedure
Description: as for outcome 14
Time Frame: 12 months
Measure: Number; unit: Participants
Arm/Group | GORE PROPATEN Vascular Graft: | Disadvantaged Autologous Vein Graft
Number analyzed (Participants) | 14 | 17
Participants
  Major Adverse Event occurred | 4 | 2
  Major Adverse Event did not occur | 10 | 15

16. Secondary Outcome: Number of Patients Surviving at One Month
Time Frame: One month
Measure: Number; unit: Participants
Arm/Group | GORE PROPATEN Vascular Graft: | Disadvantaged Autologous Vein Graft
Number analyzed (Participants) | 14 | 17
Participants
  Survived | 14 | 17
  Did not survive | 0 | 0

17. Secondary Outcome: Number of Patients Surviving at 6 Months
Time Frame: 6 months
Measure: Number; unit: Participants
Arm/Group | GORE PROPATEN Vascular Graft: | Disadvantaged Autologous Vein Graft
Number analyzed (Participants) | 14 | 17
Participants
  Survived | 13 | 16
  Did not survive | 1 | 1

18. Secondary Outcome: Number of Patients Surviving at 12 Months
Time Frame: 12 months
Measure: Number; unit: Participants
Arm/Group | GORE PROPATEN Vascular Graft: | Disadvantaged Autologous Vein Graft
Number analyzed (Participants) | 14 | 17
Participants
  Survived | 13 | 15
  Did not survive | 1 | 2

19. Secondary Outcome: Number of Patients With Wound/Graft Infection Through One Month Post-procedure
Description: Wound/graft infection was not specifically defined in the protocol and was left to the Investigator's standard of care.
Time Frame: One month
Measure: Number; unit: Participants
Arm/Group | GORE PROPATEN Vascular Graft: | Disadvantaged Autologous Vein Graft
Number analyzed (Participants) | 14 | 17
Participants
  Infected | 2 | 1
  Not infected | 12 | 16

20. Secondary Outcome: Number of Patients With Wound/Graft Infection Through 6 Months
Description: Wound/graft infection was not specifically defined in the protocol and was left to the Investigator's standard of care.
Time Frame: 6 months
Measure: Number; unit: Participants
Arm/Group | GORE PROPATEN Vascular Graft: | Disadvantaged Autologous Vein Graft
Number analyzed (Participants) | 14 | 17
Participants
  Infected | 2 | 1
  Not infected | 12 | 16

21. Secondary Outcome: Number of Patients With Wound/Graft Infection Through 12 Months
Description: Wound/graft infection was not specifically defined in the protocol and was left to the Investigator's standard of care.
Time Frame: 12 months
Measure: Number; unit: Participants
Arm/Group | GORE PROPATEN Vascular Graft: | Disadvantaged Autologous Vein Graft
Number analyzed (Participants) | 14 | 17
Participants
  Infected | 2 | 1
  Not infected | 12 | 16

22. Secondary Outcome: Number of Patients With Delayed Wound Healing Through One Month Post-procedure
Description: Delayed wound healing was not specifically defined in the protocol and was left to the Investigator's standard of care.
Time Frame: One month
Measure: Number; unit: Participants
Arm/Group | GORE PROPATEN Vascular Graft: | Disadvantaged Autologous Vein Graft
Number analyzed (Participants) | 14 | 17
Participants
  Delayed wound healing | 0 | 1
  No delayed wound healing | 14 | 16

23. Secondary Outcome: Number of Patients With Delayed Wound Healing Through 6 Months Post-procedure
Description: Delayed wound healing was not specifically defined in the protocol and was left to the Investigator's standard of care.
Time Frame: 6 months
Measure: Number; unit: Participants
Arm/Group | GORE PROPATEN Vascular Graft: | Disadvantaged Autologous Vein Graft
Number analyzed (Participants) | 14 | 17
Participants
  Delayed wound healing | 1 | 1
  No delayed wound healing | 13 | 16

24. Secondary Outcome: Number of Patients With Delayed Wound Healing Through 12 Months Post-procedure
Description: Delayed wound healing was not specifically defined in the protocol and was left to the Investigator's standard of care.
Time Frame: 12 months
Measure: Number; unit: Participants
Arm/Group | GORE PROPATEN Vascular Graft: | Disadvantaged Autologous Vein Graft
Number analyzed (Participants) | 14 | 17
Participants
  Delayed wound healing | 1 | 1
  No delayed wound healing | 13 | 16

25. Secondary Outcome: Change in Quality of Life as Evaluated by the SF-36v2® Health Survey From Baseline Through One Month Post-procedure
Description: The SF-36v2 Health Survey asks 36 questions to measure health and well-being from the patient's point of view. The responses to these questions can be presented as physical component summary and mental component summary scores. An increase in score from baseline indicates an improvement in the patient's condition and a decrease in score from baseline indicates a decline in the patient's condition. The subscale and total score ranges from 0 to 100 but is normalized so that a score of 50 is the population mean, with a standard deviation of 10.
Time Frame: One month
Population: The number of patients analyzed at 1 month does not equal the number of patients originally enrolled into the study, due to the fact that a number of enrolled patients did not have (or failed to attend) their 1 month follow-up visit prior to the termination of the study.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | GORE PROPATEN Vascular Graft: | Disadvantaged Autologous Vein Graft
Number analyzed (Participants) | 10 | 8
scores on a scale
  One month change from Baseline Mental Score | 2.9 (6.61) | 2.2 (8.77)
  One month change from Baseline Physical Score | -3.6 (8.67) | 4.4 (10.44)

ADVERSE EVENTS:
Groups:
- GORE PROPATEN Vascular Graft: GORE PROPATEN Vascular Graft
- Disadvantaged Autologous Vein Graft: Disadvantaged Autologous Vein Graft
Arm/Group | GORE PROPATEN Vascular Graft | Disadvantaged Autologous Vein Graft
Serious Adverse Events (participants affected / at risk) | 4/14 | 2/17
Other Adverse Events (participants affected / at risk) | 4/14 | 3/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GORE PROPATEN Vascular Graft (N=14) | Disadvantaged Autologous Vein Graft (N=17)
Below knee amputation (Surgical and medical procedures) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Esophageal tear (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foot amputation (Surgical and medical procedures) | 1 (1) | 0 (0)
Graft infection (Infections and infestations) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Postoperative wound infection (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Transmetatarsal amputation (Surgical and medical procedures) | 0 (0) | 1 (1)
Vascular graft occlusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GORE PROPATEN Vascular Graft (N=14) | Disadvantaged Autologous Vein Graft (N=17)
Cellulitis of leg (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Claudication (Vascular disorders) | 1 (1) | 0 (0)
Edema (General disorders) | 1 (1) | 0 (0)
Incision site erythema (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Incision site hematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Intraoperative bleeding (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Post procedural swelling (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Sepsis NOS (Infections and infestations) | 1 (1) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound healing delayed (General disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was terminated prior to completion of enrollment. The primary patency and secondary endpoints were not calculated due to the paucity of data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less